## The Chinese University of Hong Kong Faculty of Medicine The Nethersole School of Nursing

## **Consent Form**

## Effectiveness of mHealth-based survivorship programme on health-related quality of life among Vietnamese colorectal cancer survivors: A randomised controlled trial

I have thoroughly reviewed the information sheet and have been informed of the study's purpose, procedures, risks and benefits. I have had the opportunity to ask questions, and have received satisfactory replies. I understand that my participation is voluntary, and I have the right to withdraw at any time without a reason. I understand that the study involves installing Android apps on my phone, collecting personal data, and uploading it to a cloud server. Access to this data will be restricted to the IT engineer and principal investigator for research purposes. I understand that the information I provide will be used solely for this study and that my personal information will be kept confidential. I have read and understood this consent form, and I agree to participate in this study.

| Signature of Participant: | | | Date: |
|-------------------------------------------|----------------|---|-------|
| | (Printed Name: | ) | |
| Signature of Person<br>Obtaining Consent: | | | Date: |
| | (Printed Name: | ) | |